CLINICAL TRIAL: NCT01227317
Title: Prognostic Value of Novel Biomarkers in Patients With Shortness of Breath Attending an Emergency Department
Brief Title: BIOmarkers of Dyspnea IN Emergency Room
Acronym: BIODINER
Status: Completed | Type: Observational
Sponsor: ThermoFisher Scientific Brahms Biomarkers France (Industry)
Responsible Party: Sponsor
Other Study IDs: BIODINER BRAHMS France
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Severe Dyspnea; CAPD; AE COPD; Acute Heart Failure; Pulmonary Embolism
Keywords: Dyspnea; Mortality
MeSH Terms: conditions — Dyspnea; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute dyspnea in ED: Acute severe shortness of breath (SOB) in emergency Department (ED) with suspicion of acute heart failure (AHF) or Pulmonary Embolism (PE)or Community-acquired pneumonia (CAP) or acute Exacerbation of chronic obstructive pulmonary disease (AE COPD)
  Interventions: Other: Prognostic value of Biomarkers

INTERVENTIONS:
Other: Prognostic value of Biomarkers — Mr pro ADM, Mr pro ANP, PCT, Copeptin and pro endothelin value to stratify the risk in SOB patients
  Other Names: Dyspnea; Prognostic value

SUMMARY:
The purpose of this study is to evaluate the capacity of some novels biomarkers Procalcitonin (PCT), Midregional Proadrenomedullin (MR pro ADM), Midregional pro-atrial natriuretic peptide (MR pro ANP), Copeptin (CT pro arginine vasopressin), Pro endothelin to stratify the risk in severe dyspnea.

DETAILED DESCRIPTION:
In emergency department shortness of breath (SOB)is a common symptom and its cause is not easy to be identified. The risk stratifying remains a challenge, Prognostic value of biomarkers might be helpful.

ELIGIBILITY:
Inclusion Criteria:

* tachypnea > 25 /min or Pa02 < 70 mmHg or SpO2 < 93%
* diagnosis suspected: CAP, PE,EACOPD, AHF

Exclusion Criteria:

* other cause of dyspnea,
* unreachable on Day 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe acute SOB Suspicion of CAP, Acute Heart failure, AE COPD or PE
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
prognostic value of PCT, MR proADM, Mr pro ANP, Copeptin and pro endothelin in SOB | at Day 30
  all cause mortality or Intensive Care Unit(ICU) admission from inclusion to Day 30

SECONDARY OUTCOMES:
establish the diagnostic value of PCT and MR pro ANP | at admission
  Confirm the diagnostic value of PCT and it's level in sepsis and MR pro ANP in Heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Hausfater, Pr, Study Chair — ED Pitié SalpêtrièreHospital in Paris; Yann-Erick Claessens, Dr, Principal Investigator — ED Cochin Hospital in Paris; Guillaume Der Sahakian, Dr, Principal Investigator — ED Hotel Dieu Hospital in Paris; Arnaud Martinage, Dr, Principal Investigator — ED Hotel Dieu Hospital in Nantes; Fatima Rayeh, Dr, Principal Investigator — ED La Miletrie Hospital in Poitiers; Eric Weil, Pr, Principal Investigator — ED Hospital B in Lille; Luc-Marie JOLY, Dr, Principal Investigator — ED Charles Nicolle Hospital in Rouen
Locations (1):
- Emergency department of Pitié Salpetriere Hospital, Paris, Paris, France